CLINICAL TRIAL: NCT05761470
Title: A Phase II Study of Camrelizumab, Fluzoparib and Nab-paclitaxel in Neoadjuvant Therapy of Her-2 Negative Breast Cancer Patients With HRR Gene Mutation
Brief Title: Neoadjuvant Camrelizumab and Fluzoparib and Nab-paclitaxel in Early Breast Cancer With HRR Gene Mutation
Acronym: IMPARP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ying Lin (Other)
Responsible Party: Sponsor-Investigator, Ying Lin, director of department, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220430GD
Record Dates: First submitted 2022-12-24; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Her-2 Negative Breast Cancer; HRR Gene Mutation
MeSH Terms: interventions — camrelizumab; fluzoparib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Fluzoparib and Nab-paclitaxel (Experimental): Participants who confirmed pathogenic or likely pathogenic HRR gene mutation received Camrelizumab and Fluzoparib with nab-paclitaxel from the second cycle followed by nab-paclitaxel for one cycle.
  Interventions: Drug: Camrelizumab; Drug: Fluzoparib; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab at a fixed dose of 200mg via IV infusion on Days 1 each 21-day cycle.
  Fluzoparibat at a fixed dose of 100mg BID, each 21-day cycle. Nab-paclitaxel at a fixed dose of 260 milligrams via intravenous (IV) infusion on Days 1 each 21-day cycle.
Drug: Fluzoparib — Fluzoparib
Drug: Nab-paclitaxel — Nab-paclitaxel

SUMMARY:
This study is to evaluate the efficacy and safety of combination of Camrelizumab (Immunotherapy, PD-1 inhibitor), Fluzoparib (PARP inhibitor) and Nab-paclitaxel in neoadjuvant therapy of Her-2 negative breast cancer patients with HRR gene mutation.

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label phase II clinical trial investigating the activity of Camrelizumab+Fluzoparib+Nab-paclitaxel combination therapy in breast cancer patients with Her2-negative and HRR gene mutation for neoadjuvant therapy.

Anticipated 66 candidates meeting all study eligibility criteria will receive 8 cycles of Nab-paclitaxel (260mg/m2) every 3 weeks, which will add Camrelizumab (200mg, d1) and Fluzoparib (100mg BID) from the second cycle.

HRR gene mutation contains at least one pathogenic or likely pathogenic variant in germline or somatic BRCA1, BCRA2 and PALB2 genes, or in germline ATM, BARD1, BRIP1, CDK12, CHEK2, RAD51C, RAD51D genes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented Her-2 negative
* TNM stage: T1c, N1-N2；T2-4, N0-N2；any T, N3
* No distant metastatic disease
* Eastern Cooperative Oncology Group Performance Status: 0~1
* HRR gene mutation: at least one pathogenic or likely pathogenic variant in germline or somatic BRCA1, BCRA2 and PALB2 genes, or in germline ATM, BARD1, BRIP1, CDK12, CHEK2, RAD51C, RAD51D genes.

Exclusion Criteria:

* Patients who are pregnant or lactating at the time of randomization or refuse to contraception.
* Patients who have other malignant diseases within 2 years, except for cured skin basal cell carcinoma, breast carcinoma in situ or cervical carcinoma in situ
* Patients with psychiatric disorder, peripheral or central nerve system disease or any disorder, which compromises ability to give informed consent or participate in this study.
* Patients who have myocardial infarction or congestive heart failure, or other serious cardiac disease.
* Patients who have used immunosuppressive drug or corticosteroids within 14 days.
* Patients who have other diseases which researchers.
* Patients who allergy to any of the drugs in this trail.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | Up to 32 weeks
  Pathologic response will be assessed in the surgically resected cancer and lymph nodes after completion of all chemotherapy by the local pathologist as part of routine care. Pathologic complete response is defined as no invasive cancer in the resected breast tissue and lymph nodes (ypT0/Tis, ypN0).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 32 weeks
  ORR is defined as percentage of participants with Complete Response and Partial Response
Residual Cancer Burden (RCB) | Up to 32 weeks
  Pathologilly assessed residual cancer burden according to MD Anderson protocol.
Event-Free Survival (EFS) | Up to 20 years
  EFS was defined as the time from the date of randomization to the date of events from any cause.
Overall Survival (OS) | Up to 20 years
  OS was defined as the time from the date of randomization to the date of death from any cause.
Safety of drugs | Up to 32 weeks
  Adverse effects of the candidates according to NCI-CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lin, MD, Study Chair — Principal Investigator
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided